CLINICAL TRIAL: NCT03317223
Title: A Phase 3, Randomized, Double-blind, Active-controlled, Multicenter Study to Evaluate the Efficacy and Safety of a Triple Therapy With CJ-12420, Amoxicillin and Clarithromycin in H. Pylori Positive Patients
Brief Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Triple Therapy With CJ-12420 in H. Pylori Positive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJ_APA_306
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CJ-12420/Clarithromycin/Amoxicillin (Experimental): CJ-12420 50mg /Clarithromycin 500mg /Amoxicillin 1g
  Interventions: Drug: CJ-12420/Clarithromycin/Amoxicillin
- Lansoprazole/Clarithromycin/Amoxicillin (Active Comparator): Lansoprazole 30mg /Clarithromycin 500mg /Amoxicillin 1g
  Interventions: Drug: CJ-12420/Clarithromycin/Amoxicillin

INTERVENTIONS:
Drug: CJ-12420/Clarithromycin/Amoxicillin — CJ-12420 or Lansoprazole +Clarithromycin/Amoxicillin will be administrated twice a day, for 7 days
  Other Names: Lansoprazole/Clarithromycin/Amoxicillin

SUMMARY:
The current study is designed to demonstrate the non-inferiority of CJ-12420-based triple therapy (CJ-12420, amoxicillin and clarithromycin) versus lansoprazole-based triple therapy (lansoprazole, amoxicillin and clarithromycin) in H. pylori eradication rate and to evaluate the safety of CJ-12420 following oral administration of either triple therapy twice daily for 7 days in H. pylori positive patients.

DETAILED DESCRIPTION:
This is a double blind, randomized, active controlled, phase 3 study. Subjects will be randomly assigned to one of the two treatment groups (CJ-12420 50mg, lansoprazole 30mg). All subjects will be asked to take 5 tablets include clarithromycin, amoxicillin twice a day for 7 days.

After the treatment, UBT test will be conducted to confirm the Helicobacter pylori eradication.

ELIGIBILITY:
Inclusion Criteria:

* H. pylori-positive at screening
* Complain of gastric discomfort symptom

Exclusion Criteria:

* Having received prior therapy for eradication of H. pylori
* Prior use of proton pump inhibitors (PPIs), H2 receptor blockers, at a full dosage within 14 days
* Prior use of H. pylori eradication effective antibiotics, bismuth within 14 days

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
H. pylori eradication rate | twice a day
  Subjects will be considered to succeed in achieving H. pylori eradication if subject's UBT test (Eradication Assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Yong Chan Lee, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi YJ, Lee YC, Kim JM, Kim JI, Moon JS, Lim YJ, Baik GH, Son BK, Lee HL, Kim KO, Kim N, Ko KH, Jung HK, Shim KN, Chun HJ, Kim BW, Lee H, Kim JH, Chung H, Kim SG, Jang JY. Triple Therapy-Based on Tegoprazan, a New Potassium-Competitive Acid Blocker, for First-Line Treatment of Helicobacter pylori Infection: A Randomized, Double-Blind, Phase III, Clinical Trial. Gut Liver. 2022 Jul 15;16(4):535-546. doi: 10.5009/gnl220055. Epub 2022 Jul 6. PMID 35791797